CLINICAL TRIAL: NCT05449665
Title: Healthy Diets for a Healthy Weight: Exploring Physiological Mechanisms Related to Dietary Fibre
Brief Title: Focus on Fibre Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were issues with recruitment so study was stopped
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 813
Record Dates: First submitted 2022-06-17; First posted 2022-07-08 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Appetitive Behavior
Keywords: fibre; appetite control; gut microbiome; glycaemic control
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control - High Fibre - Low Fibre (CTRL - HF - LF) (Experimental): * Phase 1 - CTRL: Control diet with moderate fibre consumption for 13days.
  * Phase 2 - HF: ad libitum consumption of HF meals for 13days.
  * Phase 3 - LF: ad libitum consumption of LF meals for 13days.
  Interventions: Other: Phase 1 - Control; Other: Phase 2 - High Fibre; Other: Phase 3 - Low Fibre

INTERVENTIONS:
Other: Phase 1 - Control — Control diet (30% Fat, 15% Protein, 55% Carbohydrate, Fibre rising from 10 to 16g/d).
  Fed to energy balance (1.5 x Resting Metabolic Rate, RMR).
  Other Names: Phase 1 - CTRL
Other: Phase 2 - High Fibre — High Fibre diet (30% Fat, 15% Protein, 55% Carbohydrate, 30g/day Fibre). Fed ad libitum, contains 20g/day pectin (split over breakfast, lunch and dinner) in drinks/yoghurts which will be compulsory to consume and 10g/day fibre coming from the diet provided.
  Other Names: HF
Other: Phase 3 - Low Fibre — Low Fibre diet (30% Fat, 15% Protein, 55% Carbohydrate, 10g/day Fibre). Fed ad libitum.
  Other Names: LF

SUMMARY:
The investigators present a diet intervention study, to be conducted as a within-subject design, with all food and beverages provided, to allow ad libitum feeding to assess impact of diet change on appetite response. The diets will vary in fibre content and type. This study will allow assessment of the physiological impact of dietary fibre on markers of appetite control for body weight, measured from plasma gut hormones. The investigators propose to recruit participants with a poor diet quality (low habitual fibre intake) to additionally examine the time-course of adaptation of the gut microbiome (measured in faecal samples), whilst assessing the impact of added fibre on body weight and subjective appetite scores. This approach is to address the impact of dietary fibre in people living with obesity and food inequalities. The investigators will assess physiological bio-markers of appetite control and their contribution to the development of a gut ecosystem that promotes health. A subsequent period of return to a low fibre feeding will allow assessment of durability of response.

ELIGIBILITY:
Inclusion Criteria:

* healthy but overweight/obese (BMI 28-40kg/m2) males and females (post-menopausal, using the oral contraceptive pill or some form of hormonal contraceptive)
* low habitual fibre intake (<10g/day)

Exclusion Criteria:

Medication exclusion criteria:

* antibiotic use (within the past 3 months due to impact on gut microbiota)
* statins (current)
* aspirin or other NSAIDs or anti-coagulants (current)
* anti-depressants (current)
* smoking or vaping

Medical exclusion criteria:

* Females who are planning to be pregnant, are pregnant or are breastfeeding
* Anyone with food allergies, self-reported food sensitivity or intolerance
* Anyone with coeliac disease or gluten intolerance
* Anyone taking medication which may affect their appetite
* Anyone with an eating disorder
* Anyone with diabetes
* Anyone with a gastrointestinal disorder, kidney disease, liver disease or gout
* Anyone suffering from a psychiatric disorder or any type of substance abuse
* Anyone suffering from unregulated thyroid disease

Other exclusion criteria:

* Anyone following a vegetarian or vegan diet
* Anyone following a weight loss programme (that may be affecting lifestyle, physical activity & diet)
* Anyone with unsuitable veins for blood sampling
* Anyone who is unable to fluently speak, read and understand English
* Anyone who is unable to comply to an alcohol-free diet for 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in gut hormones to assess appetite response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by acute and chronic changes in plasma ghrelin and peptide YY (PYY)
Change in subjective hunger to assess appetite response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by acute and chronic changes in appetite using visual analogue scale questionnaires

SECONDARY OUTCOMES:
Change in gut metabolites (from faecal samples) in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by changes in faecal short chain fatty acids concentrations
Change in gut microbiome composition (from faecal samples) in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by changes in bacterial 16S ribosomal ribonucleic acid gene sequencing; 16S rRNA
Change in glycaemic control in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by acute and chronic changes in plasma glucose and insulin

OTHER OUTCOMES:
Change in blood metabolites in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by acute and chronic changes in plasma short chain fatty acids (SCFA)
Change in lipid profile in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by change in fasting plasma lipid profile (cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and non-esterified fatty acids (NEFA)
Change in diet markers in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured by change in urinary metabolites
Height | At screening visit only
  measured in metres
Change in body weight in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured as weight in kilograms
Change in blood pressure in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured as mmHg on each test day
Change in waist and hip circumferences in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  measured as in cm with a tape measure on each test day
Change in waist to hip ratio in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  waist and hip measures will be combined to report waist to hip ratio
Change in Body Mass Index (BMI) in response to dietary fibre | At baseline and end of each arm (study days 0, 14, 28 and 42)
  weight and height measures will be combined to report BMI in kg/m^2
Change in gastrointestinal symptoms in response to dietary fibre | every day of study (42days)
  measured daily, at end of day, using questionnaires
Change in appetite in response to dietary fibre | every day of study (42days)
  measured daily, at end of day, using visual analogue scale questionnaires
Change in free-living glycaemic control in response to dietary fibre | every day of study (42days)
  measured using continuous glucose monitoring (CGM)
Change in food intake | at screening (7days) and every day of study (42days)
  measured using weighed intake records

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, Prof, Principal Investigator — Rowett Institute, University of Aberdeen; Alexander Ross, Dr, Principal Investigator — Rowett Institute, University of Aberdeen
Locations (1):
- Rowett Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No